CLINICAL TRIAL: NCT00538668
Title: Radioimmunotherapy Phase I Dose-Escalation Studies in Prostate Cancer Using 177Lu-J591 Antibody: Dose Fractionation Regimen
Brief Title: Radioimmunotherapy in Prostate Cancer Using 177Lu-J591 Antibody
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0602008378; Repetitive dosing 177Lu-J591
Record Dates: First submitted 2007-10-02; First posted 2007-10-03 (Estimated); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Prostate Cancer
Keywords: Prostate; Prostate Cancer; Prostate Ca
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- 1 (Experimental): 20 mCi/m2 of 177Lu-J591 will be given in 2 doses, 2 weeks apart.
  Interventions: Drug: 117Lu-J591
- 2 (Experimental): 25 mCi/m2 of 177Lu-J591 will be given in 2 doses, 2 weeks apart.
  Interventions: Drug: 117Lu-J591
- 3 (Experimental): 30 mCi/m2 of 177Lu-J591 will be given in 2 doses, 2 weeks apart.
  Interventions: Drug: 117Lu-J591
- 4 (Experimental): 35 mCi/m2 of 177Lu-J591 will be given in 2 doses, 2 weeks apart.
  Interventions: Drug: 117Lu-J591
- 5 (Experimental): 40 mCi/m2 of 177Lu-J591 will be given in 2 doses, 2 weeks apart.
  Interventions: Drug: 117Lu-J591
- 6 (Experimental): 45 mCi/m2 of 177Lu-J591 will be given in 2 doses, 2 weeks apart.
  Interventions: Drug: 117Lu-J591
- 7 (Experimental): 50 mCi/m2 of 177Lu-J591 will be given in 2 doses, 2 weeks apart.
  Interventions: Drug: 117Lu-J591
- 8 (Experimental): 55 mCi/m2 of 177Lu-J591 will be given in 2 doses, 2 weeks apart.
  Interventions: Drug: 117Lu-J591
- 9 (Experimental): 25 mCi/m2 of 177Lu-J591 will be given every 2 weeks.
  Interventions: Drug: 117Lu-J591

INTERVENTIONS:
Drug: 117Lu-J591 — There will be 9 groups of patients. The first group will receive 20 units of test drug and the 9th group will receive 55 units of the test drug. The exact dose of the test drug will depend upon how many patients have been included in this protocol at the time of patient enrollment. Patients will receive 20-55 units (or millicuries) of radioactivity depending upon patient specific height and weight. The assignment of each patient for a specific dose level is purely based on the sequence of recruitment basis and does not depend on the clinical status of the patient.

SUMMARY:
The purpose of this study is to test the safety of the experimental drug, 177Lu-J591 and see what effects (good and bad) it has on your prostate cancer. Another purpose is to find the highest dose of the drug that can be given without causing severe side effects.

DETAILED DESCRIPTION:
Study Design: We plan to perform a phase I dose-escalation study. The trial is designed to determine the cumulative MTD in a FDR in which 177Lu-J591 will be given in 2 doses, 2 weeks apart. The dose escalation will start at 20 mCi/m2 and escalate in increments of 5 mCi/m2 to 55 mCi/m2 in up to 8 cohorts.We plan to recruit a maximum of 68 subjects in this trial.

Specific Aims: 1. Determine the cumulative MTD of 177Lu-J591 in a 2 week dose-fractionation regimen.

2. Perform imaging and pharmacokinetic (PK) studies with 177Lu-J591 in order to define the PK and dosimetry of 177Lu-J591 3. Determine the myelotoxicity of fractionated dose of 177Lu-J591 4. Monitor biochemical (PSA) and/or measurable disease response and duration.

Following the administration of 177Lu-J591 mAb on day 0, blood samples may be obtained at 10 min, 1, 2, 4 hrs, days 1, once during days 3-6, day 7 and 14. In addition, total body images may be obtained on day 0 at 1-4 hours after study treatment, day 1, once during days 3-6, days 7 and 14 using a gamma camera. (Amendment dated 15 July 2009: As investigators have gained ample information from the initial cohorts, PK and 177Lu-J591 imaging studies (other than the day 6-8 scan) will be considered optional.) Patients will be followed for a minimum of 12 weeks after the 2nd dose of 177Lu-J591 (total 14 weeks) or until toxicities resolve, disease progression or administration of alternative therapy for the patient¿s prostate cancer. Various clinical and laboratory evaluations will be performed during the first week and then every week until 12 weeks. These include, blood chemistries, CBCs, serum PSA levels, etc. If the patient¿s disease is stable or responding at 12 weeks after his last dose, he will continue to be followed until progression of disease. During the long-term follow-up, the patient¿s PSA will be monitored at least every 6 weeks and CT/bone scans will be evaluated at least every 18 weeks until disease progression.

ELIGIBILITY:
Inclusion Criteria

* Histologic diagnosis (recent or remote) of prostate adenocarcinoma
* Progressive, castrate metastatic carcinoma of the prostate defined by presence of metastatic disease on imaging and:

  * progressive tumor lesions on CT or MRI and/or
  * new osseus lesions on bone scan and/or
  * rising PSA

    * Rising PSA on 3 serial determinations over a period of greater than 2 weeks. An increase in PSA must be determined by two separate measurements taken at least one week apart and confirmed by a third and if necessary, a fourth measurement. If the third measurement is not greater than the second, then a fourth measurement must be taken. The fourth measurement must be greater than the second measurement for the patients to be eligible for enrollment in the study. The minimum final PSA must be > 2.
* For subjects who have not undergone surgical orchiectomy, LHRH agonist or antagonist therapy must me maintained for the duration of this study
* Platelet count > 150,000/mm3
* Absolute neutrophil count (ANC) ≥ 2,000/mm3
* Normal coagulation profile (defined as PT or INR and PTT < 1.3x ULN), unless on a stable anticoagulation regimen
* Hematocrit > 27% or Hemoglobin > 9 g/dL without blood transfusion dependency
* Patients of child bearing potential must agree to use an effective method of contraception
* Patient must have progressed following discontinuation of anti-androgen therapy, if received
* Serum testosterone < 50 ng/ml

Exclusion Criteria

* Prior corticosteroids and/or adrenal hormone inhibitors within 4 weeks of treatment, except for low dose maintenance prednisone or hydrocortisone (i.e. for adrenal insufficienty) on a stable dose at the investigator's discretion
* Prior cytotoxic chemotherapy and/or radiation therapy within 4 weeks of treatment.
* Prior radiation therapy encompassing >25% of expected red marrow distribution.
* Prior treatment with 89Strontium (Metastron®) or 153Samarium (Quadramet®)
* CNS metastasis
* History of seizure and/or stroke within past 6 months
* Known history of HIV
* Serum creatinine > 2x ULN
* AST > 2x ULN
* Bilirubin (total) > 1.5x ULN; subjects with Gilbert's syndrome will be allowed if direct bilirubin is within institutional normal limits
* Serious active infection (as assessed by investigator)
* Active angina pectoris or NY Heart Association Class III-IV
* ECOG Performance Status > 2
* Life expectancy < 6 months
* Age < 21 y.o
* Other serious illness(es) involving the cardiac, respiratory, CNS, renal, hepatic or hematological organ systems which might preclude completion of this study or interfere with determination of causality of any adverse effects experienced in this study
* Prior treatment with monoclonal Ab J591 labeled with therapeutic doses of 177Lu or 90Y
* Other investigational therapy within 4 weeks of treatment
* Inability to understand and the willingness to sign a written informed consent document or to follow investigational procedures in the opinion of the investigator

Ages: 21 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Define the PK and dosimetry of 177Lu-J591 | Perform imaging and pharmacokinetic (PK) sampling during the first two weeks of treatment.
Determine the cumulative maximum tolerated dose of 177Lu-J591 in a 2 week dose-fractionation regimen. | Will be determined baesd on toxicity experienced by patients at each dose level.
Determine the myelotoxicity of fractionated dose of 177Lu-J591 | Lab tests will be performed weekly.
Define the preliminary efficacy (response rate) of 177Lu-J591 | PSA will be evaluated at baseline and weeks 6, 10 and 14. Scan will be perfoemed at baseline and week 14.

SECONDARY OUTCOMES:
Monitor biochemical (PSA) and/or measurable disease response and duration. | PSA will be evaluated at baseline and weeks 6, 10 and 14. Scan will be perfoemed at baseline and week 14.
Estimate radiation dosimetry of 177Lu-J591 and correlate toxicity with radiation dosimetry. | Total body images will be obtained on day 0 at 1-4 hours after treatment, day 1, once during days 3-6, days 7 and 14

CONTACTS AND LOCATIONS:
Overall Officials: Scott Tagawa, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College-New York Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martiniova L, Zielinski RJ, Lin M, DePalatis L, Ravizzini GC. The Role of Radiolabeled Monoclonal Antibodies in Cancer Imaging and ADC Treatment. Cancer J. 2022 Nov-Dec 01;28(6):446-453. doi: 10.1097/PPO.0000000000000625. PMID 36383907
- [Derived] Vlachostergios PJ, Niaz MJ, Skafida M, Mosallaie SA, Thomas C, Christos PJ, Osborne JR, Molina AM, Nanus DM, Bander NH, Tagawa ST. Imaging expression of prostate-specific membrane antigen and response to PSMA-targeted beta-emitting radionuclide therapies in metastatic castration-resistant prostate cancer. Prostate. 2021 Apr;81(5):279-285. doi: 10.1002/pros.24104. Epub 2021 Jan 19. PMID 33465252